CLINICAL TRIAL: NCT03675009
Title: Milwaukee Day Cares Indoor Air Quality Assessment and Educational Response Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: University of Wisconsin, Milwaukee (Other)
Responsible Party: Principal Investigator, Joshua Steinberg, Assistant Professor, Medical College of Wisconsin
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Health Services Research
Other Study IDs: 5520466
Record Dates: First submitted 2018-07-10; First posted 2018-09-18 (Actual); Last update posted 2019-04-22 (Actual); Status verified 2019-04

CONDITIONS: Pollution; Exposure
Keywords: Child Day Care Centers; Indoor Air Quality; Educational Intervention

STUDY DESIGN:
Intervention Model Description: stepped wedge
Who Masked: Participant, Care Provider
Masking Description: Participants and education providers will be unaware whether they are in an early or late delivery of education randomization group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early Intervention (Other): Educational curriculum will be delivered earlier in the timeframe after IAQ monitoring has initiated.
  Interventions: Other: Educational Programming
- Late Intervention (Other): Educational curriculum will be delivered later in the timeframe after IAQ monitoring has initiated.
  Interventions: Other: Educational Programming

INTERVENTIONS:
Other: Educational Programming — Green Cleaning educational programming to day care staff.

SUMMARY:
This CTSI pilot study will assess for benefit of a community health worker or nursing student taught green cleaning curriculum (developed by the local asthma coalition) provided to Milwaukee County day care staff. Consumer grade indoor air quality monitors will be deployed before and after the educational intervention to objectively monitor changes as a result of the intervention. Surveys regarding changes in cleaning practices by day care staff will also be obtained to assess changes resulting from the intervention.

DETAILED DESCRIPTION:
A research and community service partnership of the Medical College of Wisconsin, the Univ. of Wisconsin-Milwaukee School of Nursing and the non-profit asthma coalition Fight Asthma Milwaukee Allies (FAM) was developed to describe and improve health relevant air quality conditions within urban Milwaukee daycare environments. Daycare air quality and the ability of education to improve air quality, both within Milwaukee and elsewhere, has not been extensively studied nor addressed in Wisconsin state law to date.

This project aims to understand the levels of indoor organic pollution and fine particles in the air, as well as temperature and humidity with using inexpensive, consumer-grade, internet cloud enabled continuous indoor air quality (IAQ) monitors. These air quality variables are scientifically established important risk factors for both the development and exacerbation of asthma.

This project aims to train UWM Nursing students, FAM Allies volunteers and MCW staff to teach an established educational programing curriculum developed by FAM Allies to daycare staff. Daycare programs may be motivated to participate in study as the curriculum is approved continuing education credits for daycare staff members.

The FAM Allies curriculum will address understanding of the importance of asthma and IAQ with irritant reduction measures, and safer cleaning and pest-control techniques. Additionally, the program will review the importance of IAQ upon the lungs and review knowledge about asthma.

The proposal is a 4-month intervention in which the IAQ monitor will be placed in daycares to obtain baseline measurements. Half of the facilities will receive education at the second month allowing the team to assess before and after education air quality readings. The rest of the facilities will receive the same education at the third month. After 4 months, the devices will be removed from the facilities and results in aggregate will be shared with the daycare.

ELIGIBILITY:
Inclusion Criteria:

* licensed child day care staff within Milwaukee County
* authorized consent to participate in study by day care organization

Exclusion Criteria:

* medical or adult day care centers

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-04-19 (Actual)

PRIMARY OUTCOMES:
Alterations in total Volatile Organic Compounds (tVOC) temporally associated with the educational intervention | baseline through 4 months
  Assessment of tVOC levels (ppb) before and after educational intervention, reduction an intended effect of the curriculum
Alterations in particulate matter (PM2.5) temporally associated with the educational intervention | baseline through 4 months
  Assessment of particulate matter 2.5um levels (PM2.5, ug/m3) before and after educational intervention; reduction an intended effect of the curriculum

SECONDARY OUTCOMES:
Assessment of Cleaning Practices (including VOC generation) practice changes associated with the Educational Intervention | before educational curriculum, up to 4 months following educational intervention
  Quantitative before/after surveys of Day Care cleaning behavior practices before the educational intervention and up to 4 months following, via survey inventories (practice frequencies assessed with 5 tiers survey, range: everyday to never); completed by a single designated Day Care administrator
Assessment of Perceived Obstacles to Cleaning Behavior Change | immediately following educational intervention
  Survey-based assessment of beliefs about Obstacles to Cleaning Behavior Change (ranked survey with 8 domains, scale 1-8 of importance); all child care staff participating in educational intervention
Assessment of Percieved Quality of Educational Program | immediately following educational intervention
  Survey-based assessment of beliefs about Quality of Educational Program (survey with ranked scale poor/neutral/good, 5 domains), pre-specified subgroup analysis based upon teacher type (nursing student, Americorp worker, professional asthma educator)
Baseline Description of Day Care Indoor Air Quality tVOC | period of time before educational intervention (1-2 months)
  Assessment of tVOC (ppb) averages and range before educational interventions; observed values before curriculum to establish baseline values in community, to assess if elevated values are associated with specific cleaning behaviors discouraged in the educational curriculum
Baseline Description of Day Care Indoor Air Quality PM2.5 | period of time before educational intervention (1-2 months)
  Assessment of PM2.5 (ug/m3) averages and range before educational interventions; observed values before curriculum to establish baseline values in community, to assess if elevated values are associated with specific cleaning behaviors discouraged in the educational curriculum

CONTACTS AND LOCATIONS:
Overall Officials: Anne Dressel, PhD, Principal Investigator — University of Wisconsin-Milwaukee School of Nursing; Joshua Steinberg, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-11): https://cdn.clinicaltrials.gov/large-docs/09/NCT03675009/Prot_SAP_000.pdf